CLINICAL TRIAL: NCT01057589
Title: Phase 2 Study of Pemetrexed in Combination With Cisplatin and Cetuximab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study for Patients With Recurrent or Metastatic Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12170; H3E-MC-S123 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-20; First posted 2010-01-27 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Head and Neck Neoplasms
Keywords: Pharynx; Larynx; Cervical esophagus; Nose; Thyroid Gland; Parathyroid Gland
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Thyroid Diseases | interventions — Pemetrexed; Cetuximab; Cisplatin; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Cisplatin + Cetuximab (Experimental): Participants will receive pemetrexed,cisplatin and cetuximab for up to 6 cycles (21 days per cycle) followed by optional maintenance of pemetrexed and cetuximab until disease progression. Optional maintenance therapy is permitted after at least 4 cycles of triplet combination therapy have been given. Cetuximab will be administered as an initial dose of 400 milligram per meter squared (mg/m^2) intravenous (IV) infusion and as a 250 mg/m^2 IV weekly dose thereafter.
  As Standard of care dietary supplements included: 350 to 1000 micrograms (µg) oral Folic Acid 5 times a day for the 7 days preceding the first dose of first dose of pemetrexed and continuing throughout treatment and for 21 days after the last dose of pemetrexed and 1000 µg vitamin B12 intramuscular injection (IM) during the week preceding the first dose of pemetrexed and every 9 weeks thereafter.
  Interventions: Drug: Pemetrexed; Drug: Cetuximab; Drug: Cisplatin; Dietary Supplement: Folic Acid; Dietary Supplement: Vitamin B12

INTERVENTIONS:
Drug: Pemetrexed — Triplet Combination Therapy: 500 mg/m^2 administered intravenously on Day 1 of 21 day cycle for up to 6 cycles
  Maintenance Therapy: 500mg/m^2 administered intravenously on Day 1 of 21 day cycle until disease progression or unacceptable toxicity
  Other Names: Alimta; LY231514
Drug: Cetuximab — Triplet Combination Therapy: 400 mg/m^2 administered intravenously on Day 1 of 21 day cycle for 1 cycle; 250 mg/m^2 administered IV infusion on Day 1 of 21 day cycle and then weekly for up to 6 cycles.
  Maintenance Therapy: 250 mg/m^2 administered intravenously on Day 1 of 21 day cycle and then weekly until disease progression or unacceptable toxicity
Drug: Cisplatin — Triplet Combination Therapy: 75mg/m^2 administered intravenously on Day 1 of 21 day cycle for up to 6 cycles.
Dietary Supplement: Folic Acid — Standard of care dietary supplements: 350 to 1000 µg orally 5 times a day for the 7 days preceding the first dose of first dose of pemetrexed and continuing throughout treatment and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 — Standard of care dietary supplements: 1000 µg IM during the week preceding the first dose of pemetrexed and every 9 weeks thereafter.

SUMMARY:
The purpose of this trial is to estimate progression free survival in patients with recurrent or metastatic head and neck cancer that have not received chemotherapy in this setting.

DETAILED DESCRIPTION:
A 12 patient safety lead will evaluate side effects in patients receiving at least 2 cycles of the combination pemetrexed, cisplatin and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of squamous cell carcinoma of head and neck (SCCHN)
* Recurrent or metastatic SCCHN, not amenable to local therapy
* At least 6 months since completion of systemic therapy (chemotherapy or biological anticancer therapy)
* No more than 1 prior systemic therapy, given as part of multimodal treatment for locally advanced disease;
* No prior systemic therapy for metastatic disease
* Radiation therapy must be completed at least 4 weeks before study enrollment.
* For palliative therapy, prior radiation therapy allowed to <25% of the bone marrow (Cristy and Eckerman 1987), and prior radiation to the whole pelvis is not allowed.
* Surgery (excluding prior diagnostic biopsy) must be completed at least 4 weeks before study enrollment.
* An estimated life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Oken et al. 1982).
* Biological tissue available for biomarker analysis on tumor tissue.
* Disease status may be measurable or nonmeasurable as defined by Response Evaluation Criteria in Solid Tumors
* Patient compliance and geographic proximity that allow for adequate follow-up.
* Adequate organ function
* Willingness to comply with Contraceptive Regimen
* For women: Must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen [for example, intrauterine device (IUD), birth control pills, or barrier device] during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment, and must not be breast-feeding. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period.

Exclusion Criteria:

* Nasopharyngeal, paranasal sinus, lip, or salivary gland cancer.
* Previously received treatment with monoclonal antibody therapy, or other signal transduction inhibitors of Epidermal Growth Factor Receptor therapy.
* Are receiving concurrent chronic systemic immune therapy, or chemotherapy for a disease other than cancer.
* Serious concomitant systemic disorder (for example, active infection) or psychiatric disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* Have serious cardiac disease, such as symptomatic , unstable angina, or the history of myocardial infarction in the previous 12 months.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Have had another primary malignancy other than Head and Neck cancer, unless that prior malignancy was treated at least 2 years previously with no evidence of recurrence. Exception: Patients with a history of in situ carcinoma of the cervix, nonmelanoma skin cancer, or low-grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed and treated less than 2 years previously.
* Presence of clinically significant (by physical exam) third-space fluid collections; for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
* Have peripheral neuropathy
* Have central nervous system (CNS) metastases (unless the patient has completed successful local therapy for CNS metastases and has been off corticosteroids for at least 4 weeks before starting study therapy). Brain imaging is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose less than or equal to 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Unable or unwilling to take folic acid, vitamin B12, or prophylactic corticosteroids.
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination.
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (13):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain, France
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan, Italy
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cardiff, South Glamorgan

REFERENCES:
- [Background] Cristy M, Eckerman KF. 1987. Specific absorbed fractions of energy at various ages from internal sources: I. methods. Prepared by the Oak Ridge National Laboratory, Oak Ridge, Tenn.
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Derived] Vermorken JB, Licitra L, Stohlmacher-Williams J, Dietz A, Lopez-Picazo JM, Hamid O, Hossain AM, Chang SC, Gauler TC. Phase II study of pemetrexed in combination with cisplatin and cetuximab in recurrent or metastatic squamous cell carcinoma of the head and neck. Eur J Cancer. 2013 Sep;49(13):2877-83. doi: 10.1016/j.ejca.2013.05.002. Epub 2013 May 30. PMID 23726971

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cisplatin + Cetuximab: Pemetrexed 500 milligram per meter squared (mg/m^2) administered by intravenous (IV) infusion followed by cisplatin 75 mg/m^2 administered by IV infusion both given on Day 1 of each 21 day cycle. Cetuximab 400 mg/m^2 administered by IV infusion initially as a loading dose in Week 1, subsequent weeks cetuximab 250 mg/m^2 administered by IV infusion once per week for a maximum of six 21 day cycles.
  At the discretion of the investigator participants who completed at least 4 cycles of triplet combination therapy could continue to receive pemetrexed plus cetuximab in the maintenance setting or as a monotherapy of pemetrexed or cetuximab alone in the absence of PD, unacceptable toxicity or any other withdrawal criterion up to 19 months.
  Participants also received Folic Acid and Vitamin B12 as standard of care dietary supplements.
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin + Cetuximab
Started | 66
Completed | 0
Not Completed | 66
Not completed — Disease Progression | 35
Not completed — Adverse Event | 10
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 3
Not completed — Sponsor Decision | 1
Not completed — Death | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed Cisplatin Cetuximab: Pemetrexed 500 mg/m^2 administered by IV infusion followed by cisplatin 75 mg/m^2 administered by IV infusion both given on Day 1 of each 21 day cycle. Cetuximab 400 mg/m^2 administered by IV infusion initially as a loading dose in Week 1, subsequent weeks cetuximab 250 mg/m^2 administered by IV infusion once per week for a maximum of six 21 day cycles. At the discretion of the investigator participants who completed at least 4 cycles of triplet combination therapy could continue to receive pemetrexed plus cetuximab in the maintenance setting or as a monotherapy of pemetrexed or cetuximab alone in the absence of PD, unacceptable toxicity or any other withdrawal criterion up to 19 months. Participants also received Folic Acid and Vitamin B12 as standard of care dietary supplements.
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 53
Race/Ethnicity, Customized [Number; unit: participants]
  White | 66
Region of Enrollment [Number; unit: participants]
  Belgium | 8
  France | 4
  Germany | 32
  Italy | 8
  Spain | 13
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS based on Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines defined as the time from the date of first dose of study drug to first documented objective progressive disease (PD) or death from any cause. PD is defined as at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline to date of PD or death up to 18.7 months
Population: Protocol Qualified (PQ) Population: all randomized and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 66
months | 4.4 [3.6 to 5.4]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of first dose of study drug to the date to death from any cause.
Time Frame: Baseline to date of death up to 18.7 months
Population: PQ Population: all randomized and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 66
months | 9.7 [6.5 to 13.1]

3. Secondary Outcome: Percent of Participants With a Partial Response (PR) or a Complete Response (CR)
Description: CR and PR based on RECIST Guidelines: CR is defined as the disappearance of all tumor lesions; PR is defined as at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LDs or the complete disappearance of target lesions, with persistence (but not worsening) of one or more nontarget lesions and the appearance of no new lesions. PD is defined as at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Date of first response to PD (up to 18.7 months)
Population: PQ Population: all randomized and treated participants with evaluable data; 6 participant's results were unknown.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 58
percentage of participants | 29.3 [18.1 to 42.7]

4. Secondary Outcome: Change From Baseline in Participant Reported European-Quality of Life 5 Dimension Instrument (EQ-5D) Visual Analog Scale (VAS) at End of Triplet Combination Therapy and End of Maintenance Therapy
Description: Vertical VAS - a 20 millimeter (mm), fractionated scale in the form of a thermometer with endpoints of 0 (worst imaginable health state) and 100 (best imaginable health state). Participants used the EQ-5D VAS scale to rate their overall health on the day the questionnaire was administered. Possible change values range from -100 (best imaginable health at baseline changed to worst possible health at visit) to 100 (worst possible health at baseline changed to best possible health at visit).
Time Frame: Baseline, End of Triplet Combination Therapy (up to Cycle 6 [4.2 months]), End of Maintenance Therapy (up to 18.7 months)
Population: PQ Population: all randomized and treated participants with evaluable data for each category
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 26
units on a scale
  Change at End of Triplet Therapy (n=23) | -1.2 (14.28)
  Change at End of Maintenance Therapy (n=11) | -10.6 (21.51)
Statistical Analysis 1: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.697, t-test, 2 sided — P-value is for Change at End of Triplet Combination Therapy. Threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.132, t-test, 2 sided — P-value is for Change at End of Maintenance Therapy. Threshold for statistical significance was 0.05

5. Secondary Outcome: Change From Baseline in Participant Reported EQ-5D Utility Score at End of Triplet Combination Therapy and End of Maintenance Therapy
Description: EQ-5D Index is derived by converting the Descriptive System (participant is required to rate health by checking 1 [no limitation], 2 [some limitation] or 3 [severe or complete limitation] in 5 dimensions [mobility, self-care, usual activities, pain/comfort and anxiety/depression]) to a single summary index. A utility value assigned to each individual's health state based on the absence or presence of moderate or severe problems in the 5 dimensions. A regression equation defines a utility value for these health states. The possible values for health utility ranged from -0.59 (severe problems in all 5 dimensions) to 1 (no problem in all dimensions) on a scale where 0 represents death and 1 represents the best possible health state. Possible change values range from -1.59 (no problems at baseline to severe problems at visit) to 1.59 (severe problems at baseline to no problems at visit).
Time Frame: Baseline, End of Triplet Combination Therapy (up to 6 cycles [4.2 months]) , End of Maintenance Therapy (up to 18.7 months)
Population: PQ Population: all randomized and treated participants with EQ-5D data at respective timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 34
units on a scale
  Change at End of Triplet Therapy (n=29) | 0.05 (0.230)
  Change at End of Maintenance Therapy (n=15) | -0.02 (0.291)
Statistical Analysis 1: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.223, t-test, 2 sided — P-value is for Change at End of Triplet Combination Therapy. Threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.788, t-test, 2 sided — P-value is for Change at End of Maintenance Therapy. Threshold for statistical significance was 0.05

6. Secondary Outcome: Change From Baseline in Performance Status Scale for Head and Neck Cancer Patients (PSS-HNC)
Description: PSS-HNC is a clinician-rated instrument designed to measure speaking and eating disabilities of participants with head and neck cancer and consists of 3 subscales: Normalcy of Diet (NOD) subscale measures the ability of the participants to eat a normal diet, scale ranged from 0 (non-oral feeding) to 100 (unrestricted diet); Understandability of Speech (UOS)subscale measured the degree a clinician was able to understand the participant's speech, subscale ranged from 0 (never understandable) to 100 (always understandable); Eating in Public (EIP) subscale, rating based on clinician question to the participant to report who he/she eats with and in what setting, subscale ranged from 0 (always eats alone) to 100 (no restriction of place, food, or companion). Change from baseline: negative value represents a decrease in function and a positive value represents an increase in function.
Time Frame: Baseline, Triplet Combination Therapy Cycles 2, 4, 6 (cycle = 21 days) and optional Maintenance Therapy Cycles 1, 3, 5 and 7 (cycle = 21 days)
Population: PQ Population: all randomized and treated participants with evaluable data at respective timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed Cisplatin Cetuximab
Number analyzed (Participants) | 54
units on a scale
  NOD-Change at Triplet Cycle 2 (n=53) | -0.4 (20.8)
  NOD-Change at Triplet Cycle 4 (n=41) | 3.9 (24.2)
  NOD-Change at Triplet Cycle 6 (n=24) | 3.3 (23.5)
  NOD-Change at Maintenance Cycle 1 (n=23) | 0.4 (29.9)
  NOD-Change at Maintenance Cycle 3 (n=10) | -1.0 (21.3)
  NOD-Change at Maintenance Cycle 5 (n=6) | 8.3 (20.4)
  NOD-Change at Maintenance Cycle 7 (n=5) | -8.0 (11.0)
  EIP-Change at Triplet Cycle 2 (n=46) | 2.7 (25.4)
  EIP-Change at Triplet Cycle 4 (n=37) | -6.8 (29.3)
  EIP-Change at Triplet Cycle 6 (n=22) | -3.4 (20.8)
  EIP-Change at Maintenance Cycle 1 (n=23) | -8.7 (38.1)
  EIP-Change at Maintenance Cycle 3 (n=10) | -10.0 (21.1)
  EIP-Change at Maintenance Cycle 5 (n=6) | -4.2 (24.6)
  EIP-Change at Maintenance Cycle 7 (n=5) | -15.0 (22.4)
  UOS-Change at Triplet Cycle 2 (n=53) | 0.5 (18.0)
  UOS-Change at Triplet Cycle 4 (n=41) | -4.3 (17.6)
  UOS-Change at Triplet Cycle 6 (n=24) | -10.4 (22.0)
  UOS-Change at Maintenance Cycle 1 (n=23) | -1.1 (14.1)
  UOS-Change at Maintenance Cycle 3 (n=10) | -2.5 (7.9)
  UOS-Change at Maintenance Cycle 5 (n=6) | -12.5 (34.5)
  UOS-Change at Maintenance Cycle 7 (n=5) | -15.0 (33.5)
Statistical Analysis 1: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.90, t-test, 2 sided — P-value is for NOD, Triplicate Combination Therapy Cycle 2. Threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.31, t-test, 2 sided — P-value is for NOD, Triplicate Combination Therapy Cycle 4. Threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.49, t-test, 2 sided — P-value is for NOD, Triplicate Combination Therapy Cycle 6. Threshold for statistical significance was 0.05
Statistical Analysis 4: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.95, t-test, 2 sided — P-value is for NOD, Maintenance Cycle 1. Threshold for statistical significance was 0.05
Statistical Analysis 5: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.89, t-test, 2 sided — P-value is for NOD, Maintenance Cycle 3. Threshold for statistical significance was 0.05
Statistical Analysis 6: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.36, t-test, 2 sided — P-value is for NOD, Maintenance Cycle 5. Threshold for statistical significance was 0.05
Statistical Analysis 7: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.18, t-test, 2 sided — P-value is for NOD, Maintenance Cycle 7. Threshold for statistical significance was 0.05
Statistical Analysis 8: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.47, t-test, 2 sided — P-value is for EIP, Triplicate Combination Cycle 2. Threshold for statistical significance was 0.05
Statistical Analysis 9: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.17, t-test, 2 sided — P-value is for EIP, Triplicate Combination Cycle 4. Threshold for statistical significance was 0.05
Statistical Analysis 10: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.45, t-test, 2 sided — P-value is for EIP, Triplicate Combination Cycle 6. Threshold for statistical significance was 0.05
Statistical Analysis 11: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — P-value is for EIP, Maintenance Cycle 1. Threshold for statistical significance was 0.05
Statistical Analysis 12: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.17, t-test, 2 sided — P-value is for EIP, Maintenance Cycle 3. Threshold for statistical significance was 0.05
Statistical Analysis 13: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.70, t-test, 2 sided — P-value is for EIP, Maintenance Cycle 5. Threshold for statistical significance was 0.05
Statistical Analysis 14: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.21, t-test, 2 sided — P-value is for EIP, Maintenance Cycle 7. Threshold for statistical significance was 0.05
Statistical Analysis 15: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.85, t-test, 2 sided — P-value is for UOS, Triplicate Combination Cycle 2. Threshold for statistical significance was 0.05
Statistical Analysis 16: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.13, t-test, 2 sided — P-value is for UOS, Triplicate Combination Cycle 4. Threshold for statistical significance was 0.05
Statistical Analysis 17: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.03, t-test, 2 sided — P-value is for UOS, Triplicate Combination Cycle 6. Threshold for statistical significance was 0.05
Statistical Analysis 18: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.71, t-test, 2 sided — P-value is for UOS, Maintenance Cycle 1. Threshold for statistical significance was 0.05
Statistical Analysis 19: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.34, t-test, 2 sided — P-value is for UOS, Maintenance Cycle 3. Threshold for statistical significance was 0.05
Statistical Analysis 20: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.41, t-test, 2 sided — P-value is for UOS, Maintenance Cycle 5. Threshold for statistical significance was 0.05
Statistical Analysis 21: Comparison: Pemetrexed Cisplatin Cetuximab; Test type: Superiority or Other; p = 0.37, t-test, 2 sided — P-value is for UOS, Maintenance Cycle 7. Threshold for statistical significance was 0.05

ADVERSE EVENTS:
Arm/Group | Pemetrexed Cisplatin Cetuximab
Serious Adverse Events (participants affected / at risk) | 45/66
Other Adverse Events (participants affected / at risk) | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Cisplatin Cetuximab (N=66)
Anaemia (Blood and lymphatic system disorders) | 4 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Asthenia (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 2 (2)
Implant site haemorrhage (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Medical device pain (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2)
Performance status decreased (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (4)
Anaphylactic shock (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (4)
Sepsis (Infections and infestations) | 2 (2)
Septic embolus (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asterixis (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Cisplatin Cetuximab (N=66)
Anaemia (Blood and lymphatic system disorders) | 26 (30)
Leukopenia (Blood and lymphatic system disorders) | 26 (36)
Neutropenia (Blood and lymphatic system disorders) | 26 (35)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (19)
Conjunctivitis (Eye disorders) | 6 (7)
Lacrimation increased (Eye disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 25 (29)
Diarrhoea (Gastrointestinal disorders) | 20 (28)
Dyspepsia (Gastrointestinal disorders) | 10 (11)
Dysphagia (Gastrointestinal disorders) | 12 (13)
Nausea (Gastrointestinal disorders) | 27 (33)
Stomatitis (Gastrointestinal disorders) | 20 (24)
Vomiting (Gastrointestinal disorders) | 22 (26)
Asthenia (General disorders) | 14 (25)
Chills (General disorders) | 4 (4)
Fatigue (General disorders) | 40 (45)
Mucosal inflammation (General disorders) | 22 (35)
Oedema peripheral (General disorders) | 7 (9)
Pain (General disorders) | 4 (5)
Pyrexia (General disorders) | 12 (12)
Folliculitis (Infections and infestations) | 6 (6)
Oral candidiasis (Infections and infestations) | 4 (5)
Creatinine renal clearance decreased (Investigations) | 4 (4)
Weight decreased (Investigations) | 10 (10)
Weight increased (Investigations) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 29 (31)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Fluid retention (Metabolism and nutrition disorders) | 6 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (26)
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 (24)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Dizziness (Nervous system disorders) | 15 (18)
Dysgeusia (Nervous system disorders) | 7 (8)
Neuropathy peripheral (Nervous system disorders) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Acne (Skin and subcutaneous tissue disorders) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (12)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (17)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 31 (37)
Skin fissures (Skin and subcutaneous tissue disorders) | 11 (12)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4)
Hypotension (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days